CLINICAL TRIAL: NCT03604627
Title: Study of Coronary Calcium Score as a Marker of Post-radiation Vascular Dysplasia in Adults Treated During Childhood for Cancer With Mediastinal Irradiation
Acronym: COROCAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-A02256-47; 2017/2610 (Other: CSET number)
Record Dates: First submitted 2018-07-20; First posted 2018-07-27 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Childhood Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated for cancer during childhood or adolescence (Other): Patients over the age of 18 treated during childhood or adolescence for cancer with irradiation affecting the heart area (≥20% of ≥5Gy heart volume) and / or anthracyclines (≥ 300mg/m^²)
  Interventions: Other: Coronal calcium score measurement

INTERVENTIONS:
Other: Coronal calcium score measurement — A medical interview with clinical examination by a cardiologist for screening cardiovascular risk factors, including smoking, and looking for symptoms of heart disease as part of routine care.
  In accordance with routine care, a fasting and fasting blood test will be performed performed on exam day at Bichat Hospital or at another time, close to the patient's home according to his availability. The biological blood test will include the measurement of plasma triglyceride concentrations, total cholesterol and its HDL and LDL fractions, blood glucose, glycated hemoglobin and serum creatinine with estimated glomerular filtration rate according to the CKD-EPI formula. Sample urinalysis will include measurement of creatinine, proteinuria, and microalbuminuria.
  An electrocardiogram (ECG) rest, a cardiac ultrasound, a test and respiratory function tests (EFR) will be performed as part of routine care. Coronal calcium score measurement will be performed as part of the research.

SUMMARY:
To measure coronary calcium score in adults treated during childhood or adolescence for irradiation cancer in the heart and / or anthracycline area and compare them to determine whether irradiation of the heart area is associated with increased calcium score after adjustment for other cardiovascular risk factors (age, sex, smoking, dyslipidemia, obesity, diabetes, high blood pressure and renal failure).

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older,
2. Treated for cancer during childhood, adolescence or young adulthood (≤25 years),
3. Treated with irradiation of the heart area (≥20% of ≥5Gy heart rate) and / or anthracycline (cumulative dose of doxorubicin equivalent ≥300mg/m^²),
4. In complete remission of their pediatric cancer for at least 10 years,
5. Patient affiliated to a social security scheme or beneficiary of such a scheme,
6. Patient Information and Signed Informed Consent.

Exclusion Criteria:

1. Perspective less than 10 years,
2. Persons deprived of liberty or guardianship (including trusteeship),
3. Impossibility of submitting to the medical follow-up of the test for geographical, social or psychological reasons,
4. Pregnant women.

Inclusion criteria for extension cohort:

1. Patients 30 years of age or older,
2. Treated for cancer during childhood, adolescence or young adulthood (≤25 years),
3. Treated with irradiation of the heart area (≥20% of ≥5Gy heart rate),
4. In complete remission of their pediatric cancer for at least 10 years,
5. Patient affiliated to a social security scheme or beneficiary of such a scheme,
6. Patient Information and Signed Informed Consent.

Exclusion criteria for extension cohort:

1. Persons deprived of liberty or guardianship (including trusteeship),
2. Impossibility of submitting to the medical follow-up of the test for geographical, social or psychological reasons,
3. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-06-14 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of a calcium score | Up to 24 months
  Incidence of a calcium score measured by the Agatston score> 0 in the study population of adults treated during childhood or adolescence for cancer with irradiation of the heart area and / or treatment with anthracyclines

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Gustave Roussy, Villejuif, Val De Marne
  - Hôpital Bichat, Paris
  - Hôpital Trousseau, Paris

IPD SHARING:
Plan to Share IPD: No